CLINICAL TRIAL: NCT03725033
Title: Multicentre Double-blind Placebo-controlled Parallel Group Randomized Clinical Trial of Efficacy and Safety of Subetta in the Treatment of Impaired Glucose Tolerance
Brief Title: Clinical Trial of Efficacy and Safety of Subetta in the Treatment of Impaired Glucose Tolerance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-SU-006
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Results first posted 2021-01-14 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2019-11

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — subetta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subetta (Experimental): Tablet for oral use. 2 tablets twice daily. The tablets should be held in mouth until completely dissolved 15 min prior to meal.
  Interventions: Drug: Subetta
- Placebo (Placebo Comparator): Tablet for oral use. 2 tablets twice daily. The tablets should be held in mouth until completely dissolved 15 min prior to meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Subetta — Oral administration.
  Arms: Subetta
Drug: Placebo — Oral administration.
  Arms: Placebo

SUMMARY:
Purpose of the study:

* to assess the efficacy of Subetta in the treatment of impaired glucose tolerance
* to assess the safety of Subetta in the treatment of impaired glucose tolerance.

DETAILED DESCRIPTION:
Design: a multicenter, double-blind, placebo-controlled, parallel-group randomized trial.

The study will enroll outpatients adults aged 18 to 70 years with impaired glucose tolerance (IGT) who did not receive glucose-lowering agents previously. Persons with pre-diabetes, obesity (especially with visceral or abdominal obesity), dyslipidemia (with high triglycerides and/or low-density lipoproteins), hypertension, diabetes in first-degree relatives will be considered as potential candidates to participate in the study.

After the patient's information sheet and the form of informed consent for participation in the study are signed on the screening (visit 0; day from -7 to 0), complaints and history are collected, registration of concomitant conditions and diseases, objective examination, calculation of body mass index (BMI), oral glucose tolerance test (OGTT), fasting blood glucose. Furthermore, blood samples (for testing HbA1c, chemistry and hematology, HLA genotyping) and urine sample will be collected; concomitant therapy will be recorded, diet and physical activity recommendations will be given. All women of childbearing potential will be administered pregnancy tests.

If eligibility criteria are met and there are no non-inclusion criteria on Visit 1 (Day 1), the patient is randomized to one of two groups: the Subetta group (patients will take 2 tablets twice a day for 12 weeks) or placebo group (patients will take a placebo according to the scheme of Subetta for 12 weeks).

In the course of the study, two more visits in 4 (Visit 2) and 12 (Visit 3) weeks are planned, during these weeks complaints are recorded, a patient's examination is recorded, therapy compliance and safety are assessed. On Visit 3 OGTT, fasting blood glucose, blood samples (for HbA1c, chemistry and hematology) and urinalysis will be performed.

The duration of observation period shall be up to 13 weeks. During the study the treatment for underlying conditions will be allowed with the exception of the drugs indicated in the section "Prohibited concomitant therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients aged 18 to 70 years.
2. Impaired glucose tolerance (plasma glucose from 7.8 to 11.0 mmol / L 2 hours after a 75 g oral glucose consumption during an oral glucose tolerance test, while fasting plasma glucose <7.0 mmol / L).
3. HbA1c is 5.7-6.4%.
4. The body mass index is 25.0-39.9 kg / m^2.
5. Consent to use reliable contraceptive methods during the study (for men and women with reproductive potential).
6. The presence of the signed informed consent form to participate in the clinical trial.

Exclusion Criteria:

1. Type 1 or type 2 diabetes.
2. Use of any medications indicated in the section "Prohibited concomitant medications".
3. Acute or exacerbation / decompensation of a chronic disease of any etiology at the time of the examination or during the previous week.
4. Uncontrolled arterial hypertension with blood pressure: systolic blood pressure > 160 mm Hg and/or diastolic blood pressure > 110 mm Hg.
5. Acute coronary syndrome, myocardial infarction, acute impairment of cerebral circulation during the previous 6 months prior to enrollment.
6. Unstable or life-threatening arrhythmia during the previous 3 months prior to enrollment.
7. Acute and chronic heart failure with functional class III or IV (according to the classification of the New York Heart Association, 1964).
8. Respiratory failure.
9. Chronic kidney disease (classes C3-5 A3).
10. Hepatic insufficiency (class C according to Child-Pugh).
11. Presence or suspicion of oncology disease.
12. The presence of an allergy / hypersensitivity to any component of the medication administered during the treatment.
13. Alcohol consumption > 2 alcohol units for males and > 1 alcohol unit for females per day.
14. Mental illness or drug abuse in anamnesis.
15. Bariatric surgery in anamnesis, any surgery for 3 months before enrollment.
16. Pregnancy, breast-feeding; childbirth less than 3 months before enrollment.
17. Participation in other clinical trials for 3 months before enrollment in this study.
18. Patients who are related to any of the on-site research personnel directly involved in the conduct of the trial or are an immediate relative of the study investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
19. Patients who work for MATERIA MEDICA HOLDING (i.e. the company's employees, temporary contract workers, appointed officials responsible for carrying out the research or immediate relatives of the aforementioned).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- Russia (44):
  - Arkhangelsk Regional Clinical Hospital, Arkhangelsk
  - Belgorod State National Research University, Belgorod
  - Kirov Clinical Hospital № 7 named. V.I. Yurlova, Kirov
  - Kuban State Medical University, Krasnodar
  - Regional Clinical Hospital #1 named after Professor Ochapovsky, Krasnodar
  - Clinic of Professor Gorbakov, Krasnogorsk
  - Krasnogorsk city hospital №1, Krasnogorsk
  - City Clinical Hospital named after F.I. Inozemtseva Department of Health of Moscow, Moscow
  - City Clinical Hospital named after V.P. Demikhova, Moscow
  - Moscow Clinical Scientific and Practical Center of the Moscow City Health Department, Moscow
  - The Federal State Budgetary Healthcare Institution The Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - Pirogov Russian National Research Medical University, Moscow
  - Federal State Institution "Polyclinic No. 5" of the Administrative Department of the President of the Russian Federation, Moscow
  - National Medical Research Center for Rehabilitation and Balneology, Moscow
  - LLC Clinic "Bessalar", Moscow
  - Moscow State University of Medicine and Dentistry, Moscow
  - City Clinical Hospital No. 10 of the Kanavinsky District of Nizhny Novgorod, Nizhny Novgorod
  - Semashko Nizhny Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - LLC "Medical Center "Healthy Family", Novosibirsk
  - Institute of Cytology and Genetics of the Siberian Branch of the Russian Academy of Sciences, Novosibirsk
  - Novosibirsk State Medical University, Novosibirsk
  - Rostov State Medical University, Rostov-on-Don
  - Polyclinic Complex JSC, Saint Petersburg
  - City Clinical Hospital #109, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 25", Saint Petersburg
  - Federal State Budget Military Educational Institution of Higher Education "Military Medical Academy named after S.M. Kirov Defense Ministry of the RF/Department and clinic of field therapy, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 117", Saint Petersburg
  - St. Petersburg State Budgetary Institution of Health "City Polyclinic № 54", Saint Petersburg
  - Road Clinical Hospital JSC Russian Railways, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Limited Liability Company Gastroenterologichesky Center Expert, Saint Petersburg
  - St. Petersburg State Budgetary Institution of Health "City Polyclinic № 106", Saint Petersburg
  - Pokrovskaya City Hospital, Saint Petersburg
  - St. Petersburg State Budgetary Institution of Health "City Polyclinic №4", Saint Petersburg
  - Samara city hospital #4, Samara
  - LLC Center "Diabetes", Samara
  - Saratov State Medical University named after V. I. Razumovsky, Saratov
  - Volgograd State Medical University, Volgograd
  - Voronezh Regional Clinical Consultative and Diagnostic Center, Voronezh
  - LLC "Medical Consultations and Research Center - PRACTICE", Yaroslavl
  - The State Budgetary Healthcare Institution of the Yaroslavl Region "Regional Clinical Hospital", Yaroslavl
  - Ural State Medical University, Yekaterinburg
  - City Clinical Hospital #40, Yekaterinburg
  - Central City Hospital #7, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening procedures 336 patients were excluded by the researchers because they did not meet the inclusion criteria, or they had non-inclusion criteria.
Period: Overall Study
Arm/Group | Subetta | Placebo
Started | 105 | 97
Completed | 105 | 97
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subetta: Oral administration. 2 tablets 2 times a day 15 minutes before meals. Keep the tablets in your mouth, not swallowing, until completely they are dissolved.
  Subetta: For oral use.
- Placebo: Oral administration. 2 tablets 2 times a day 15 minutes before meals. Keep the tablets in your mouth, not swallowing, until completely they are dissolved.
  Placebo: For oral use.
- Total: Total of all reporting groups
Arm/Group | Subetta | Placebo | Total
Number analyzed (Participants) | 105 | 97 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.3) | 56.1 (8.6) | 56.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 75 | 153
  Male | 27 | 22 | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 105 | 97 | 202

OUTCOME MEASURES:

1. Primary Outcome: Change 2-hour Plasma Glucose (During Oral Glucose Tolerance Test).
Description: Based on medical records. For oral glucose tolerance test, the subject is given 75 g of oral glucose and blood sample is taken 2 hours later. All analysis will be done in a central laboratory.
Time Frame: At baseline and after 12 weeks of treatment.
Population: 9 randomized patients who received full treatment and underwent all procedures according to the protocol (n = 4, Subetta group; n = 5, Placebo group) were excluded from analysis. Blood samples were obtained but the central laboratory did not provide carbohydrate metabolism values due to technical reasons for these patients.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 101 | 92
mmol/L
  Baseline | 9.27 (0.88) | 9.11 (0.86)
  After 12 weeks | 7.28 (2.07) | 8.32 (2.44)
  ∆ between baseline and after 12 weeks | -1.99 (2.21) | -0.79 (2.55)
Statistical Analysis 1: Comparison: Subetta vs Placebo; This analysis applies to ∆ between baseline and after 12 weeks row; Test type: Superiority; p = 0.0028, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percentage of Patients With 2-hour Plasma Glucose <7.8 mmol / L.
Description: Based on medical records.
Time Frame: After 12 weeks of treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 101 | 92
Participants | 64 | 46
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.0805, Fisher Exact

3. Secondary Outcome: Change in Fasting Plasma Glucose.
Description: Based on medical records. Fasting plasma glucose is measured after fasting or not eating anything for at least 8 hours.
Time Frame: At baseline and after 12 weeks of treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 101 | 92
mmol/L
  Baseline | 5.83 (0.62) | 5.88 (0.60)
  After 12 weeks | 6.01 (1.17) | 6.02 (0.92)
  ∆ between baseline and after 12 weeks | 0.18 (1.25) | 0.14 (1.06)
Statistical Analysis 1: Comparison: Subetta vs Placebo; This analysis applies to ∆ between baseline and after 12 weeks row; Test type: Superiority; p = 0.99, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in HbA1c
Description: Based on medical records. HbA1c is determined by the method certified in accordance with National Glycohemoglobin Standardization Program and standardized in compliance with the reference values adopted in the Diabetes Control and Complications Trial.
Time Frame: At baseline and after 12 weeks of treatment.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 101 | 92
percentage of HbA1c
  Baseline | 5.9 [5.8 to 6.1] | 6.0 [5.85 to 6.2]
  After 12 weeks | 5.8 [5.5 to 6.0] | 5.9 [5.6 to 6.05]
  ∆ between baseline and after 12 weeks | -0.1 [-0.5 to -0.1] | -0.1 [-0.4 to -0.1]
Statistical Analysis 1: Comparison: Subetta vs Placebo; This analysis applies to ∆ between baseline and after 12 weeks row; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the study - 12 weeks.
Arm/Group | Subetta | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/97
Other Adverse Events (participants affected / at risk) | 15/105 | 20/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subetta (N=105) | Placebo (N=97)
Pain in the abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1) — Pain in the upper abdomen (in the hypochondrium)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Acute respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Acute bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Acute conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Acute cystitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Increase of leukocytes in the urine (Investigations) | 1 (1) | 0 (0)
Increase of alanine aminotransferase levels (Investigations) | 1 (1) | 1 (1)
Increase of aspartate aminotransferase level (Investigations) | 0 (0) | 1 (1)
Increase of glycated hemoglobin level (Investigations) | 0 (0) | 1 (1)
Increase of blood pressure (Investigations) | 1 (1) | 3 (3)
Weight loss (Investigations) | 1 (1) | 1 (1)
Postprandial hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Nasal bleeding
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Knee pain
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Deterioration of the condition (General disorders) | 1 (1) | 0 (0)
Unsteadiness of gait (General disorders) | 1 (1) | 0 (0)
Concussion of the brain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Contusion of the soft tissues of the right thigh

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03725033/Prot_SAP_000.pdf